CLINICAL TRIAL: NCT03676270
Title: Trends in Modern Phase 1 Oncology Trials
Acronym: Phase 1
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB-2018Phase I
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Cancer
Keywords: Cancer; Phase I trials; Review
MeSH Terms: conditions — Neoplasms | interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Phase I — Chemotherapy, ITK, Hormotherapy, Immunotherapy

SUMMARY:
Overview of response rate published in recent oncology phase I trials

DETAILED DESCRIPTION:
Critics have raised a fundamental ethical challenge about phase 1 cancer research. They point to an expected paucity of benefits, since approximately 5% of patients in phase 1 trials are reported to have tumor shrinkage.

Objective was to conduct a search of the literature using PubMed to identify articles about phase 1 trials that were published from January 1, 2014, through June 30, 2015. The primary end point was the response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

Clinically relevant trials' characteristics were investigated as candidate factors associated with the RR: Funding source (Academic / Industrial), First-in man trial (Yes / No), Expansion cohort (Yes / No), Number of targeted organs (Single / Multiple), Therapy (Single / Combination), Treatment (MAB-Immuno / ITK / Chimioth-HT-other), Biological eligibility criterion (Yes / No), as well as the number of assessable patients, which for ease of clinical interpretation was transformed into a qualitative variable (0-25 / 26 - 50 / 51+).

The RR was described according to the individual trials' characteristics. Associations with trials's characteristics were investigated using statistical modeling.

ELIGIBILITY:
Trials based on the following eligibility criteria:

* cancer phase 1 trials
* published from January 1, 2014, through June 30, 2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unit of analysis = trial (analysis of aggregated data only, with the trial as the unit of analysis)
Sampling Method: Non-Probability Sample
Enrollment: 6915 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, MD-PhD, Principal Investigator — Institut Bergonié
Locations (1):
- Insitut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chakiba C, Grellety T, Bellera C, Italiano A. Encouraging Trends in Modern Phase 1 Oncology Trials. N Engl J Med. 2018 Jun 7;378(23):2242-2243. doi: 10.1056/NEJMc1803837. No abstract available. PMID 29874526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 224 trials were analyzed which included 6915 participants
Units Other Than Participants: trials
Groups:
- Participants Included in Phase 1 Oncology Trials: Participants included in Phase 1 Oncology Trials, published from January 1, 2014, through June 30, 2015.
Period: Overall Study
Arm/Group | Participants Included in Phase 1 Oncology Trials
Started | 6915; 224 trials
Completed | 6915; 224 trials
Not Completed | 0; 0 trials

BASELINE CHARACTERISTICS:
Groups:
- Trials: Cancer Phase 1 trials
Arm/Group | Trials
Number analyzed (Participants) | 6915
Age, Customized [Count of Participants; unit: Participants]
  trials with participant > 18 years old | 6915
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3458
  Male | 3457
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Number of reported responses (complete [CR] and partial [PR]) divided by the number of reported assessable patients
Time Frame: up to 6 months after treatment initiation
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Oncology Trials: Phase 1 Oncology Trials, published from January 1, 2014, through June 30, 2015.
Arm/Group | Phase 1 Oncology Trials
Number analyzed (Participants) | 6915
Participants | 1371

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Participants Included in Phase 1 Oncology Trials
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes